CLINICAL TRIAL: NCT01427283
Title: A Randomized, Double-blind, Double-dummy, Placebo-controlled, Active-controlled, Parallel-group, Multicenter Trial of Oxycodone/Naloxone Controlled-release Tablets (OXN) to Assess the Analgesic Efficacy (Compared to Placebo) and the Management of Opioid-induced Constipation (Compared to Oxycodone Controlled-release Tablets (OXY)) in Opioid-experienced Subjects With Moderate to Severe Chronic Low Back Pain and a History of Opioid-induced Constipation Who Require Around-the-clock Opioid Therapy
Brief Title: A Study of Oxycodone/Naloxone Controlled-release Tablets (OXN) to Assess Analgesic Efficacy and Management of Opioid-induced Constipation (OIC) in Opioid-experienced Subjects With Moderate to Severe Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONU3705; 2011-005061-20 (EudraCT Number)
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Low Back Pain
Keywords: Low back pain; Chronic pain; Opioid; Constipation; Moderate to severe
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Constipation | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- OXN (Experimental): Oxycodone/Naloxone controlled-release tablets (OXN)
  Interventions: Drug: Oxycodone/Naloxone controlled-release
- OXY (Active Comparator): Oxycodone HCl controlled-release tablets (OXY)
  Interventions: Drug: Oxycodone HCl controlled-release
- Placebo (Placebo Comparator): Placebo tablets to match OXN or OXY
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxycodone/Naloxone controlled-release — Oxycodone/Naloxone controlled-release tablets (10/5 - 40/20 mg) taken orally every 12 hours
  Arms: OXN
Drug: Oxycodone HCl controlled-release — Oxycodone HCl controlled-release tablets (10 - 40 mg) taken orally every 12 hours
  Other Names: OxyContin
  Arms: OXY
Drug: Placebo — Placebo tablets to match OXN or OXY taken orally every 12 hours
  Arms: Placebo

SUMMARY:
The primary objective is to assess the efficacy of oxycodone/naloxone controlled-release tablets (OXN) for the management of opioid-induced constipation (OIC) compared with oxycodone controlled-release tablets (OXY) in subjects with moderate to severe low back pain and opioid-induced constipation who require around-the-clock opioid therapy.

ELIGIBILITY:
Inclusion Criteria include:

* Male and female subjects ≥ 18 years of age with moderate to severe, chronic low back pain (lasting at least several hours daily) as their predominant pain condition for at least 3 months prior to screening period;
* The low back pain must be related to nonmalignant and nonneuropathic conditions and may be with or without radiation;
* Subjects must have a self-reported history of opioid induced constipation (OIC).

Exclusion Criteria include:

* Subjects with rheumatoid arthritis or other inflammatory arthritis;
* Subjects with neuropathic conditions that have been painful or required therapy within the past 3 months;
* Subjects with evidence of significant structural abnormalities of the gastrointestinal (GI) tract or other significant conditions affecting GI motility;
* Subjects with chronic constipation not related to opioid use;
* Subjects who had surgical procedures directed towards the source of chronic low back pain within 6 months of the screening visit or planned during the study;
* Subjects with a history of malignancy within past 2 years, with exception of basal cell carcinoma that has been successfully treated.

Other protocol specific inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2011-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Overall complete spontaneous bowel movement (CSBM) responder rates | Weeks 1 through 12
  The overall Complete Spontaneous Bowel Movement (CSBM) responder rates over the 12 week double-blind period comparing OXN to OXY

SECONDARY OUTCOMES:
CSBM Responder at least 50% of the weeks in the double-blind period | Weeks 1 through 12
Laxative-free Responder at least 50% of the weeks in the double-blind period | Weeks 1 through 12

CONTACTS AND LOCATIONS:
Locations (117):
- United States (117):
  - Investigational Site, Alabaster, Alabama
  - Investigational Site, Birmingham, Alabama
  - Investigational Site, Foley, Alabama
  - Investigational Site, Mobile, Alabama
  - Investigational Site, Mesa, Arizona
  - Investigational Site, Phoenix, Arizona
  - Investigational Site, Sun Lakes, Arizona
  - Investigational Site, Tucson, Arizona
  - Investigational Site, Little Rock, Arkansas
  - Investigational Site, Sherwood, Arkansas
  - Investigational Site, Anaheim, California
  - Investigational Site, Artesia, California
  - Investigational Site, Cerritos, California
  - Investigational Site, Chino, California
  - Investigational Site, El Cajon, California
  - Investigational Site, Encino, California
  - Investigational Site, Fountain Valley, California
  - Investigational Site, Fresno, California
  - Investigational Site, Garden Grove, California
  - Investigational Site, Laguna Hills, California
  - Investigational Site, Lakewood, California
  - Investigational Site, Lincoln, California
  - Investigational Site, Lomita, California
  - Investigational Site, Long Beach, California
  - Investigational Site, Oceanside, California
  - Investigational Site, Orange, California
  - Investigational Site, Paramount, California
  - Investigational Site, Sacramento, California
  - Investigational Site, San Bernardino, California
  - Investigational Site, San Diego, California
  - Investigational Site, Thousand Oaks, California
  - Investigational Site, Torrance, California
  - Investigational Site, Colorado Springs, Colorado
  - Investigational Site, Denver, Colorado
  - Investigational Site, Golden, Colorado
  - Investigational Site, Aventura, Florida
  - Investigational Site, Bradenton, Florida
  - Investigational Site, Chiefland, Florida
  - Investigational Site, Clermont, Florida
  - Investigational Site, Daytona Beach, Florida
  - Investigational Site, DeLand, Florida
  - Investigational Site, Edgewater, Florida
  - Investigational Site, Fort Lauderdale, Florida
  - Investigational Site, Fort Myers, Florida
  - Investigational Site, Hialeah, Florida
  - Investigational Site, Inverness, Florida
  - Investigational Site, Jacksonville, Florida
  - Investigational Site, Miami, Florida
  - Investigational Site, Miami Beach, Florida
  - Investigational Site, Naples, Florida
  - Investigational Site, New Smyrna Beach, Florida
  - Investigational Site, North Miami, Florida
  - Investigational Site, Oldsmar, Florida
  - Investigational Site, Orlando, Florida
  - Investigational Site, Oviedo, Florida
  - Investigational Site, Plantation, Florida
  - Investigational Site, Tamarac, Florida
  - Investigational Site, Tampa, Florida
  - Investigational Site, West Palm Beach, Florida
  - Investigational Site, Atlanta, Georgia
  - Investigational Site, Austell, Georgia
  - Investigational Site, Snellville, Georgia
  - Investigational Site, Boise, Idaho
  - Investigational Site, Chicago, Illinois
  - Investigational Site, Evansville, Indiana
  - Investigational Site, Indianapolis, Indiana
  - Investigational Site, Michigan City, Indiana
  - Investigational Site, Wichita, Kansas
  - Investigational Site, Edgewood, Kentucky
  - Investigational Site, Lake Charles, Louisiana
  - Investigational Site, Monroe, Louisiana
  - Investigational Site, New Orleans, Louisiana
  - Investigational Site, Pikesville, Maryland
  - Investigational Site, Brockton, Massachusetts
  - Investigational Site, Worcester, Massachusetts
  - Investigational Site, Florissant, Missouri
  - Investigational Site, Las Vegas, Nevada
  - Investigational Site, Atco, New Jersey
  - Investigational Site, Great Neck, New York
  - Investigational Site, Kew Gardens, New York
  - Investigational Site, New York, New York
  - Investigational Site, Rochester, New York
  - Investigational Site, Williamsville, New York
  - Investigational Site, Durham, North Carolina
  - Investigational Site, Elkin, North Carolina
  - Investigational Site, High Point, North Carolina
  - Investigational Site, Winston-Salem, North Carolina
  - Investigational Site, Columbus, Ohio
  - Investigational Site, Dayton, Ohio
  - Investigational Site, Moraine, Ohio
  - Investigational Site, Toledo, Ohio
  - Investigational Site, Oklahoma City, Oklahoma
  - Investigational Site, Eugene, Oregon
  - Investigational Site, Jenkintown, Pennsylvania
  - Investigational Site, Levittown, Pennsylvania
  - Investigational Site, Mechanicsburg, Pennsylvania
  - Investigational Site, Pittsburgh, Pennsylvania
  - Investigational Site, Red Lion, Pennsylvania
  - Investigational Site, State College, Pennsylvania
  - Investigational Site, Warwick, Rhode Island
  - Investigational Site, Charleston, South Carolina
  - Investigational Site, Myrtle Beach, South Carolina
  - Investigational Site, Rapid City, South Dakota
  - Investigational Site, Jackson, Tennessee
  - Investigational Site, Allen, Texas
  - Investigational Site, Austin, Texas
  - Investigational Site, Dallas, Texas
  - Investigational Site, Houston, Texas
  - Investigational Site, McKinney, Texas
  - Investigational Site, North Richland Hills, Texas
  - Investigational Site, Tomball, Texas
  - Investigational Site, Orem, Utah
  - Investigational Site, Salt Lake City, Utah
  - Investigational Site, Danville, Virginia
  - Investigational Site, Midlothian, Virginia
  - Investigational Site, Richmond, Virginia
  - Investigational Site, Bothell, Washington